CLINICAL TRIAL: NCT03021785
Title: A Multi-center, Open-label Phase I Study to Evaluate the Safety, Pharmacokinetics and Preliminary Efficacy of Multiple Intravitreal Injection TK001 in Patients With Neovascular Age-Related Macular Degeneration
Brief Title: A Study of Multiple Intravitreal Injection TK001 in Patients With Neovascular Age-related Macular Degeneration
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu T-Mab Biopharma Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tmab-TK001-AMD-02
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Neovascular Age-Related Macular Degeneration
Keywords: Neovascular Age-Related Macular Degeneration; Anti-VEGF; CNV; TK001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0.5mg (Experimental): In the core study, patients will receive 0.5mg TK001 in a 50-μL solution administered as an intravitreal injection every 4 weeks. In the extension study, they will be evaluated every 4 weeks and administrated PRN (pro re nata) with their assigned dose.
  Interventions: Biological: TK001
- 1.0mg (Experimental): In the core study, patients will receive 1.0mg TK001 in a 50-μL solution administered as an intravitreal injection every 4 weeks. In the extension study, they will be evaluated every 4 weeks and administrated PRN (pro re nata) with their assigned dose.
  Interventions: Biological: TK001
- 1.5mg (Experimental): In the core study, patients will receive 1.5mg TK001 in a 50-μL solution administered as an intravitreal injection every 4 weeks. In the extension study, they will be evaluated every 4 weeks and administrated PRN (pro re nata) with their assigned dose.
  Interventions: Biological: TK001

INTERVENTIONS:
Biological: TK001 — TK001 will be administered intravitreal injection.
  Other Names: anti-VEGF humanized monoclonal antibody injection

SUMMARY:
This is a multicenter, open-label study to evaluate the safety, pharmacokinetics, immunogenicity, and preliminary efficacy of multiple intravitreal injection TK001 in patients with AMD. It consists of core study (12 weeks) and extension study (40 weeks).

DETAILED DESCRIPTION:
This is a multicenter, open-label study to evaluate the safety, pharmacokinetics, immunogenicity, and preliminary efficacy of multiple intravitreal injection TK001 in patients with AMD. It consists of core study (12 weeks) and extension study (40 weeks). In the core study, patients will receive their assigned dose in a 50-μL solution administered as an intravitreal injection every 4 weeks. In the extension study, they will be evaluated every 4 weeks and administrated PRN (pro re nata) with their assigned dose. The safety, pharmacokinetics, immunogenicity, and preliminary efficacy of TK001 will be evaluated in the core study, and will also be assessed in the extension study except pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Aged 45 - 80 years, male or female
* Diagnosed with neovascular AMD and with active lesions
* Best corrected VA for the studied eye≤20/40
* With stable blood pressure, SBP<140 mmHg and DBP<90 mmHg

Exclusion Criteria:

Limitation of eye diseases

* With vitreous hemorrhage in studied eyes within two months preceding screening
* With geographic atrophy, epiretinal membrane or intensive subfoveal hard exudates which involved the foveal in studied eyes
* With opacity of refractive media(e.g. apparent cataract) or contraction of pupils which significantly interfered the visual test or assessment of anterior segment and fundus in studied eyes
* With pseudoexfoliation syndrome, intraocular hemorrhage resulting in decreased vision, rhegmatogenous retinal detachment, macular hole or choroidal neovascularization (CNV) for any reason except for AMD (such as fundus angioid streaks, ocular histoplasmosis, pathologic myopia, trauma) in studied eyes
* With apparent afferent pupillary defect(APD) in studied eyes
* With Polypoidal Choroidal Vasculopathy (PCV) or Retinal Angiomatous Proliferation (PAP) in studied eyes
* With intraocular pressure higher than 25mmHg despite treatment
* With VA for the fellow eyes<20/200
* With active inflammation in any eye, such as conjunctivitis, keratitis, scleritis, blepharitis, endophthalmitis and uveitis The treatment of the eye
* The studied eye received topical or grid photocoagulation more than twice or within 3 months preceding screening
* The studied eye received the following intraocular surgery or laser treatment in macular (such as macular translocation surgery, glaucoma filtering surgery, transpupillary thermotherapy, macular photocoagulation, vitreous cutting surgery, optic nerve dissection, optic nerve sheath membrane dissection). But patients who received verteporfin photodynamic therapy, cataract surgery or YAG posterior capsular dissection more than 3 months before screening will not be excluded.
* Any eye received antiangiogenic drugs within 2 months preceding screening or patients received systemic antiangiogenic drugs within 3 months preceding screening (such as pegaptanib, aflibercept, ranibizumab, bevacizumab or conbercept)
* Any eye received intraocular injection of corticosteroid drugs (such as triamcinolone acetonide) within 3 months preceding screening, or periocular injection of corticosteroid drugs within 1 month before screening Systemic diseases, treatment and other conditions
* With a history of allergy to sodium fluorescein and indocyanine green
* PLT≤100×109/L, BUN or Cr>1.5×ULN(Upper Limit of Normal), TT(thrombin time) or PT(prothrombin time) >1.0×ULN(Upper Limit of Normal), take anti-platelet aggregation drugs or anticoagulants within 1 month before screening
* With surgery within 1 month before screening, or with unhealed wound, ulcer, fracture at present
* Diabetic patients without the control of glucose or accompanied by diabetic retinopathy
* With a history of myocardial infarction within 6 months before screening
* With activity disseminated intravascular coagulation and a tendency of significant bleeding before screening
* Systemic autoimmune disease
* Any uncontrolled diseases (such as severe systemic diseases of mental, neurological, cardiovascular, respiratory and malignancies)
* Pregnant and lactating women or patients who cannot take contraceptive measures
* Poor compliance
* Patients who participated other clinical trials within 30 days before screening or was taking other clinical trials at present
* Patients who is considered unsuitable for enrollment by investigator

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-10-18 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Frequency of ocular and systemic AEs (adverse events) and SAEs (serious adverse events) which are related to TK001 in the first 12 weeks | 12 weeks
  Core Study
Frequency of ocular and systemic AEs (adverse events) and SAEs (serious adverse events) which are related to TK001 in the following 40 weeks | 40 weeks
  Extension Study

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) | 12 weeks
  Core Study
Maximum plasma concentration (Cmax) | 12 weeks
  Core Study
Time to reach maximum concentration (Tmax) | 12 weeks
  Core Study
Elimination half-Life (T½) | 12 weeks
  Core Study
Change from baseline in the Best Corrected Visual Acuity at 12 weeks | 12 weeks
  Core Study
Change from baseline in the mean central retinal thickness at 12 weeks | 12 weeks
  Core Study
Change from baseline in the thickness of choroidal neovascularization at 12 weeks | 12 weeks
  Core Study
Change from baseline in the retinal thickness in the site of lesion which was the thickest at 12 weeks | 12 weeks
  Core Study
Change from baseline in macular volume at 12 weeks | 12 weeks
  Core Study
Change from baseline in the area of choroidal neovascularization at 12 weeks | 12 weeks
  Core Study
Change from baseline in the area of leakage at 12 weeks | 12 weeks
  Core Study
Change from baseline in the total lesion size at 12 weeks | 12 weeks
  Core Study
Percentage of Participants Positive for anti-TK001 antibody at 12 weeks | 12 weeks
  Core Study
Change from baseline in the Best Corrected Visual Acuity at 52 weeks | 40 weeks
  Extension Study
Change from baseline in the mean central retinal thickness at 52 weeks | 40 weeks
  Extension Study
Change from baseline in the thickness of choroidal neovascularization at 52 weeks | 40 weeks
  Extension Study
Change from baseline in the retinal thickness in the site of lesion which was the thickest at 52 weeks | 40 weeks
  Extension Study
Change from baseline in macular volume at 52 weeks | 40 weeks
  Extension Study
Change from baseline in the area of choroidal neovascularization at 52 weeks | 40 weeks
  Extension Study
Change from baseline in the area of leakage at 52 weeks | 40 weeks
  Extension Study
Change from baseline in the total lesion size at 52 weeks | 40 weeks
  Extension Study
Percentage of Participants Positive for anti-TK001 antibody at 52 weeks | 40 weeks
  Extension Study

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhang, Principal Investigator — West China Hospital
Locations (5):
- China (5):
  - Chinese Academy of Medicine Sciences，Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Henan Province People's Hospital, Zhengzhou, Henan
  - ShangHai General Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The Eye Hospital of WMU(Zhejiang eye hospital), Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided